CLINICAL TRIAL: NCT00209898
Title: Hepatitis C Treatment of Inmates. A Randomized, Open-label Study Evaluating the Feasibility, Safety and Efficacy of Treatment With Peginterferon Alfa-2a in Combination With Ribavirin in Inmate Patients With Chronic Hepatitis C
Brief Title: Hepatitis C Treatment of Inmates
Acronym: PEGPRI
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low inclusion rate
Sponsor: Haukeland University Hospital (Other)
Collaborators: Bergen Prison, Norwegian Correctional Service (Other); Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Steinar Skrede, Consultant, Haukeland University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12952
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2003-06

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatits C; peginterferon; ribavirin; inmate; fast initiation procedure
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rapid standard of care (Active Comparator): Rapid standard of care treatment after screening
  Interventions: Procedure: Fast initiation procedure
- Ordinary standard of care (Active Comparator): Subject put on ordinary waiting list for hcv treatment in Our outpatient clinic
  Interventions: Procedure: Fast initiation procedure

INTERVENTIONS:
Procedure: Fast initiation procedure

SUMMARY:
Hepatitis C infection is a prevalent chronic disease. It is particularly prevalent among intravenous drug abusers. Bergen fengsel is a regional prison housing 250 inmates, of which as many as 70 are recorded HCV RNA PCR positive annuallly. In this study inmate males and females will be randomized to standard screening and initiation procedure, or to a rapid initiation procedure in the hospital's infectious diseases outpatient clinic. The study aims at studying if rapid inclusion will increase the possibility to conclude treatment while the prisoner still is incarcerated, thus improve the chances of reaching a sustained virologic response, compared to standard inclusion, where prisoners, as other out patients will wait for inclusion for several months.

ELIGIBILITY:
Inclusion Criteria:

* Serologic evidence of chronic hepatitis C infection by an anti-HCV test
* Serum HCV-RNA quantifiable at > 600 IU/mL or 1000 copies/mL by the Roche AMPLICOR HCV MONITOR Test, v2.0
* Patients with both normal or elevated serum ALT are eligible
* Compensated liver disease (Child-Pugh grade A clinical classification)
* Patients with cirrhosis or transition to cirrhosis must have an abdominal ultrasonography, CT scan or MRI scan without evidence of hepatocellular carcinoma and a serum AFP < 100 ng/mL within 2 months of randomization
* Negative urine or blood pregnancy test (for women of childbearing potential) documented within the 24 hour period prior to first dose of study drug
* All fertile males and females receiving RBV must be using two forms of effective contraception during treatment and during the 6 months after treatment ends

Exclusion Criteria:

* Women with ongoing pregnancy or breat feeding
* Therapy with any systemic anti-viral, anti-neoplastic or immunomodulatory treatment (including supraphysiologic soses of steroids and radiation) < 6 months prior to the first dose of study drug
* Any investigational drug < 6 weeks prior to the first dose of study drug Positive test at screening for anti-HAV IgM Ab, HBsAg, anti-HBsAg, anti-HBc Ab, anti-HIV Ab.
* History or evidence of a medical condition associated with chronic liver disease other than HCV (e.g. hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
* History or evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease
* Neutrophil count < 1500/mm or platelet count < 90,000 cells/mm at screening
* Serum creatinine level > 1,5 times the ULN at screening
* History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or neuroleptica at therapeutic doses for major depression or psychosis, respectively for at least 3 months at any previous time, or any history of the following; a suicidal attempt, hospitalization for psychiatric disease or a period of disability due to psychiatric disease
* History of severe seizure disorder or current anticonvulsant disease
* History of immunologically mediated disease (e.g. IBD, ITP, LED, AIHA, scleroderma, severe psoriasis or RA etc.)
* History or other evidence of chronic pulmonary disease associated with functional limitation
* History of major organ transplantation with an existing functional graft
* History of severe cardiac disease (e.g. NYHA Functional Class III or IV, myocardial infarction within 6 months of ventricular arrhythmias requiring ongoing treatment, unstable angina or other significant CVD)
* History or other evidence of severe illness, malignancy or other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* Evidence of severe retinopathy (e.g. CMV retinitis, macula degeneration)
* Evidence of ongoing drug abuse (including excessive alcohol consumption)
* Inability or unwillingness to provide informed consent or abide by the requirements of the study
* Male partners of women who are pregnant
* Hemoglobin < 12 g/dL in women or < 13g/dL in men at screening
* Any patient with an increased baseline risk for anemia or for whom anemia would be medically problematic
* Patients with documented or presumed coronary artery disease or cerebrovascular disease should not be enrolled if, in the judgement of the investigator, an acuter decrease in hemoglobin by up to 4 g/dL would not be well-tolerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2003-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
- adherence
- Sustained virologic response rates defined as percentage of patients with non-detectable HCV-RNA as measured by Roche AMPLICOR HCV Test, v2.0 (>50 IU/mL).

SECONDARY OUTCOMES:
Percentage of patients with non-detectable HCV-RNA at study week 12, 24 and 48 as measured by Roche AMPLICOR HCV Test v2.0 (<50 IU/mL).
- adverse event rate and profile
- Hemoglobin
- Other laboratory tests
- Medical Outcomes Study 36 Item Short Form health Survey (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Steinar Skrede, M.D., Ph.D., Principal Investigator — Unit for infectious diseases, Dept. Internal Medicine, Haukeland UH
Locations (1):
- Unit for infectious diseases outpatient clincic, Dept. Internal Medicine, Bergen, Bergen, Norway

REFERENCES:
- [Background] -Dalgard,O., Jeansson, S., Skaug, K, Raknerud, N., Bell, H. Hepatitis C in the general adult population of Oslo; prevalence and clinical spectrum. Scand. J. Gastroenterol. 38:864-870, 2003. -Stein, M.D., Maksad, J., Clarke, J. Hepatitis C among injecting drug users: knowledge, perceived risk and willingness to receive treatment. Drug Alc. Depend. 61:211-215, 2001. -Allen,S.A., Spaulding,A.C., Osei,A.M., Taylor,L.E., Cabral,A.M. and Rich,J.D. Treatment of chronic hepatitis C in a state correctional facility. Ann. Intern. Med. 138:187-190, 2003. -Dalgard,O., Bjøro,K., Hellum,K., Skaug,K., Gutigard,B.,Bell, H. Treatment of chronic hepatitis C in injecting drug users: 5 years' folow up. Eur. Addict. Res. 8:45-49, 2002.